CLINICAL TRIAL: NCT04273061
Title: Canadian Atezolizumab Precision Targeting for Immunotherapy Intervention
Brief Title: Investigating the Effects of Atezolizumab in People Whose Tumour DNA or RNA Indicates Possible Sensitivity
Acronym: CAPTIV-8
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-04010
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Lung Cancer; Gastrointestinal Cancer; Genitourinary Cancer; Gynecologic Cancer; Sarcoma; Unknown Primary Tumors; Head and Neck Cancer; Skin Cancer
Keywords: Genomic analysis; Atezolizumab; Whole genome and transcriptome analysis; Immune Burden Variant score; Immune checkpoint inhibition; Personalized OncoGenomics; Phase 2; Precision targeting
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms; Urogenital Neoplasms; Sarcoma; Neoplasms, Unknown Primary; Head and Neck Neoplasms; Skin Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Intervention Model Description: Simon 2-stage design; 8 tumour-defined cohorts consisting of 8 to 24 participants each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Breast Cohort (Experimental): Cohort of participants whose primary tumour type is breast.
  Interventions: Drug: Atezolizumab
- Lung Cohort (Experimental): Cohort of participants whose primary tumour type is lung.
  Interventions: Drug: Atezolizumab
- GI Cohort (Experimental): Cohort of participants whose primary tumour type is gastrointestinal (including pancreas and hepatobiliary).
  Interventions: Drug: Atezolizumab
- GU Cohort (Experimental): Cohort of participants whose primary tumour type is genitourinary.
  Interventions: Drug: Atezolizumab
- Gyne Cohort (Experimental): Cohort of participants whose primary tumour type is gynecological.
  Interventions: Drug: Atezolizumab
- Sarcoma Cohort (Experimental): Cohort of participants whose primary tumour type is sarcoma.
  Interventions: Drug: Atezolizumab
- Primary Unknown Cohort (Experimental): Cohort of participants whose primary tumour type is unknown.
  Interventions: Drug: Atezolizumab
- Other Cohort (Experimental): Cohort of participants whose primary tumour type is not classified as one of the other study arms. This cohort includes participants with cancers from the head and neck, skin, or rare cancers.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg by intravenous infusion every 3 weeks as tolerated
  Other Names: TECENTRIQ

SUMMARY:
This study will investigate the effects of atezolizumab on select cancer types in people whose analysis of tumour DNA and RNA indicates they may be sensitive to atezolizumab. This study aims to determine if the information from the cancer genome analysis corresponds with the effects of atezolizumab on individuals and their cancer.

This is a Phase 2 study, which is undertaken after preliminary safety testing on a drug is completed, and will involve approximately 200 participants. Participants are assigned to one of 8 cohorts based on their primary tumour type: breast, lung, gastrointestinal (GI), primary unknown, genitourinary (GU), sarcoma, gynecological, and 'other' cancer types. Participants in all cohorts will receive the same dose of atezolizumab (1200 mg every 3 weeks). In the first stage for each cohort, 8 participants will be enrolled and if no participants respond to treatment, enrollment to that cohort will be closed. If 1 or more participants respond to treatment, up to 16 additional participants will be enrolled to that cohort. Participants continue on treatment until they no longer may benefit from the treatment or they decide to stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years at the time of signature of informed consent.
* Participants with an incurable solid tumour who have undergone whole genome and transcriptome analysis (WGTA) as part of Personalized OncoGenomics (POG) or equivalent program.

  a. Participants must have had successful sequencing of their tumour, been formally reviewed by the POG (or POG-approved) genome analysts and found to have CAPTIV-8 factors identified (including Immune, Burden, Variant (IBV) score ≥ 5), been reviewed at the Molecular Tumour Board (MTB) (or site equivalent), and allocated to a specific tumour-defined cohort (that is open for enrolment) with a final opinion documented.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Participants must have measurable disease, as defined by RECIST 1.1.
* Life expectancy of at least 12 weeks.
* Adequate hematologic and end-organ function, as defined by the following laboratory results obtained within 28 days prior to the first study treatment:

  1. Absolute neutrophil count (ANC) ≥ 1500 cells/µL without granulocyte colony- stimulating factor support.
  2. White blood cell (WBC) counts > 2500/µL.
  3. Lymphocyte count ≥ 500/µL.
  4. Serum albumin ≥ 2.5 g/dL.
  5. Platelet count ≥ 100,000/µL without transfusion (without transfusion within 2 weeks of laboratory test used to determine eligibility).
  6. Hemoglobin ≥ 9.0 g/dL, participants may be transfused or receive erythropoietic treatment to meet this criterion.
  7. International normalized ratio (INR) or activated partial thromboplastin time (aPTT) ≤ 1.5 × Upper Limit of Normal (ULN). This applies only to participants who are not receiving therapeutic anticoagulation; participants receiving therapeutic anticoagulation must have an INR or aPTT within therapeutic limits for at least 1 week prior to enrolment.
  8. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 × ULN with the following exceptions: i) Participants with documented liver metastases: AST and/or ALT ≤ 5 × ULN. ii) Participants with documented liver or bone metastases: ALP ≤ 5 × ULN.
  9. Serum bilirubin ≤ 1.5 × ULN. Participants with known Gilbert's syndrome who have serum bilirubin level ≤ 3 × ULN may be enrolled.
  10. Serum creatinine ≤ 1.5 × ULN.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of less than 1% (one percent) per year during the treatment period and for at least 5 months after the last dose of atezolizumab.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse with a female partner of childbearing potential or who is pregnant) or use contraceptive measures that result in a failure rate of less than 1% (one percent) per year, and agreement to refrain from donating sperm, during the treatment period and for at least 5 months after the last dose of atezolizumab.
* Asymptomatic participants with treated or untreated CNS lesions are eligible provided that all of the following criteria are met:

  1. Measurable disease, per RECIST 1.1, must be present.
  2. The participant has no history of intracranial hemorrhage or spinal cord hemorrhage.
  3. The participant has not undergone stereotactic radiotherapy within 7 days prior to the initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
  4. The participant has no ongoing requirement for corticosteroids as therapy for CNS disease. Anticonvulsant therapy at a stable dose is permitted.
* Ability to give informed consent for the study procedures defined in this protocol.

Exclusion Criteria:

* Any prior treatment with monoclonal antibodies targeting the Programmed Death 1/Ligand (PD-1/PD-L1) axis, including antibody-drug conjugates and other experimental agents.
* Treatment with any approved or investigational agent or participation in another clinical trial with therapeutic intent within 14 days or five half-lives of the drug, whichever is longer, prior to enrollment. Participants receiving gonadotropin releasing hormone (GnRH) analogues may continue to receive treatment while participating in CAPTIV-8.
* Pregnancy or breastfeeding.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation.
* Active autoimmune disease at any point within the last 2 years prior to enrollment including but not limited to:

  1. Myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.
  2. Participants with a history of autoimmune-related hypothyroidism on a stable dose of thyroid-replacement hormone may be eligible for this study.
  3. Participants with controlled Type I diabetes mellitus on a stable dose of insulin regimen are eligible for this study.
* Participants with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., participants with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  1. Rash must cover less than 10% (ten percent) of body surface area (BSA).
  2. Disease is well controlled at baseline and only requiring low potency topical steroids.
  3. No acute exacerbations of underlying condition within the last 12 months requiring treatment with either psoralen plus ultraviolet radiation (PUVA), methotrexate, retinoids, biologic agents, oral calcineurin inhibitors or high potency or oral steroids.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Positive test for HIV (participants with a history of/or symptoms of HIV are eligible only if serological tests are negative).
* Participants with hepatitis B virus (HBV) are excluded if one of the following conditions is met:

  1. Positive hepatitis B surface antigen (HBsAg) test at screening; or
  2. Negative or positive hepatitis B surface antibody (HBsAb) test at screening accompanied by a positive total hepatitis B core antibody (HBcAb) test followed by a positive (per local laboratory definition) HBV DNA test.
* Positive hepatitis C virus (HCV) antibody test followed by a positive HCV RNA test at screening.
* Active tuberculosis.
* Severe infections within 2 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina.
* Major surgical procedure within 21 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study.
* Prior allogeneic stem cell or solid organ transplant.
* Treatment with systemic immunostimulatory agents (including but not limited to interferons, interleukin-2 (IL-2)) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to Cycle 1, Day 1.
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1, or anticipated requirement for systemic immunosuppressive medications during the trial.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
* Participants who are otherwise felt by the treating clinician to be unfit to proceed with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) in each tumour-defined cohort, as defined by RECIST 1.1 | From the date of the screening scan (within 28 days of first dose) until the date of confirmed progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  The proportion of participants in each tumour-defined cohort who have a complete response (CR) or partial response (PR) to treatment, as defined by RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) in each tumour-defined cohort from the initiation of atezolizumab | From the date of first dose until the date of confirmed progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  The length of time from the first dose of atezolizumab until participants in each tumour-defined cohort have progressive disease (PD), as defined by RECIST 1.1.
Clinical benefit rate (CBR) in each tumour-defined cohort at the 18-week follow-up scan | From the date of the screening scan (within 28 days of first dose) until the date of the 18-week follow-up scan.
  The percentage of participants in each tumour-defined cohort who have a complete response (CR), partial response (PR), or stable disease (SD) response to treatment, as defined by RECIST 1.1, at the 18-week follow-up scan.
Overall survival (OS) in each tumour-defined cohort from the initiation of atezolizumab | From the date of first dose until the date of death, assessed up to 54 months.
  The length of time from the initiation of atezolizumab that participants in each tumour-defined cohort survive.
Quality-adjusted survival in each tumour-defined cohort from the initiation of atezolizumab | From the date of first dose until the treatment discontinuation visit (within 30 days of last dose), withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  Survival time (from the initiation of atezolizumab) multiplied by quality of life. Participants' responses to health-related quality of life questions on the EQ-5D-3L questionnaire will be converted to utility weights using existing conversion scales that are based on patient and public valuations of the health states described by the EQ-5D-3L questionnaire.
Duration of response (DoR) in each tumour-defined cohort | From the date of the scan that shows the first response to treatment until the date of progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  The length of time from the first response to treatment (CR or PR) until participants in each tumour-defined cohort have progressive disease (PD), as defined by RECIST 1.1.

OTHER OUTCOMES:
Putative markers of sensitivity to atezolizumab in each tumour-defined cohort | From the date of screening sample collection until the date of progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  From blood and tissue samples collected throughout the study, identify putative markers of sensitivity to atezolizumab based on the response to treatment of the participants in each tumour-defined cohort.
Putative primary and secondary resistance markers to atezolizumab in each tumour-defined cohort | From the date of screening sample collection until the date of progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  From blood and tissue samples collected throughout the study, identify putative primary and secondary resistance markers to atezolizumab based on the response to treatment of the participants in each tumour-defined cohort.
Putative germline predictors of adverse events or toxicities of interest in each tumour-defined cohort | From the date of screening sample collection until the date of progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  From blood and tissue samples collected throughout the study, identify putative germline predictors of adverse events or toxicities of interest to atezolizumab based on the response to treatment of the participants in each tumour-defined cohort.
Compare the utility of iRECIST for response assessment to RECIST 1.1 in each tumour-defined cohort | From the date of the screening scan (within 28 days of first dose) until the date of progression, withdrawal, or date of death, whichever comes first, assessed up to 54 months.
  Participant response to treatment as per RECIST 1.1. compared to the response to treatment as per the modified response evaluation criteria in solid tumours for immunotherapy trials (iRECIST) from screening until progression in each tumour-defined cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Janessa Laskin, MD, Principal Investigator — BC Cancer
Locations (2):
- Canada (2):
  - BC Cancer, Vancouver, British Columbia
  - University Health Network / Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ayers M, Lunceford J, Nebozhyn M, Murphy E, Loboda A, Kaufman DR, Albright A, Cheng JD, Kang SP, Shankaran V, Piha-Paul SA, Yearley J, Seiwert TY, Ribas A, McClanahan TK. IFN-gamma-related mRNA profile predicts clinical response to PD-1 blockade. J Clin Invest. 2017 Aug 1;127(8):2930-2940. doi: 10.1172/JCI91190. Epub 2017 Jun 26. PMID 28650338
- [Background] Balachandran VP, Luksza M, Zhao JN, Makarov V, Moral JA, Remark R, Herbst B, Askan G, Bhanot U, Senbabaoglu Y, Wells DK, Cary CIO, Grbovic-Huezo O, Attiyeh M, Medina B, Zhang J, Loo J, Saglimbeni J, Abu-Akeel M, Zappasodi R, Riaz N, Smoragiewicz M, Kelley ZL, Basturk O; Australian Pancreatic Cancer Genome Initiative; Garvan Institute of Medical Research; Prince of Wales Hospital; Royal North Shore Hospital; University of Glasgow; St Vincent's Hospital; QIMR Berghofer Medical Research Institute; University of Melbourne, Centre for Cancer Research; University of Queensland, Institute for Molecular Bioscience; Bankstown Hospital; Liverpool Hospital; Royal Prince Alfred Hospital, Chris O'Brien Lifehouse; Westmead Hospital; Fremantle Hospital; St John of God Healthcare; Royal Adelaide Hospital; Flinders Medical Centre; Envoi Pathology; Princess Alexandria Hospital; Austin Hospital; Johns Hopkins Medical Institutes; ARC-Net Centre for Applied Research on Cancer; Gonen M, Levine AJ, Allen PJ, Fearon DT, Merad M, Gnjatic S, Iacobuzio-Donahue CA, Wolchok JD, DeMatteo RP, Chan TA, Greenbaum BD, Merghoub T, Leach SD. Identification of unique neoantigen qualities in long-term survivors of pancreatic cancer. Nature. 2017 Nov 23;551(7681):512-516. doi: 10.1038/nature24462. Epub 2017 Nov 8. PMID 29132146
- [Background] Bolotin DA, Shugay M, Mamedov IZ, Putintseva EV, Turchaninova MA, Zvyagin IV, Britanova OV, Chudakov DM. MiTCR: software for T-cell receptor sequencing data analysis. Nat Methods. 2013 Sep;10(9):813-4. doi: 10.1038/nmeth.2555. Epub 2013 Jul 28. No abstract available. PMID 23892897
- [Background] Bolotin DA, Poslavsky S, Mitrophanov I, Shugay M, Mamedov IZ, Putintseva EV, Chudakov DM. MiXCR: software for comprehensive adaptive immunity profiling. Nat Methods. 2015 May;12(5):380-1. doi: 10.1038/nmeth.3364. No abstract available. PMID 25924071
- [Background] Brown SD, Warren RL, Gibb EA, Martin SD, Spinelli JJ, Nelson BH, Holt RA. Neo-antigens predicted by tumor genome meta-analysis correlate with increased patient survival. Genome Res. 2014 May;24(5):743-50. doi: 10.1101/gr.165985.113. Epub 2014 Apr 29. PMID 24782321
- [Background] Brown SD, Raeburn LA, Holt RA. Profiling tissue-resident T cell repertoires by RNA sequencing. Genome Med. 2015 Nov 30;7:125. doi: 10.1186/s13073-015-0248-x. PMID 26620832
- [Background] Cibulskis K, Lawrence MS, Carter SL, Sivachenko A, Jaffe D, Sougnez C, Gabriel S, Meyerson M, Lander ES, Getz G. Sensitive detection of somatic point mutations in impure and heterogeneous cancer samples. Nat Biotechnol. 2013 Mar;31(3):213-9. doi: 10.1038/nbt.2514. Epub 2013 Feb 10. PMID 23396013
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Freeman JD, Warren RL, Webb JR, Nelson BH, Holt RA. Profiling the T-cell receptor beta-chain repertoire by massively parallel sequencing. Genome Res. 2009 Oct;19(10):1817-24. doi: 10.1101/gr.092924.109. Epub 2009 Jun 18. PMID 19541912
- [Background] Gogvadze E, Buzdin A. Retroelements and their impact on genome evolution and functioning. Cell Mol Life Sci. 2009 Dec;66(23):3727-42. doi: 10.1007/s00018-009-0107-2. Epub 2009 Aug 2. PMID 19649766
- [Background] Hugo W, Zaretsky JM, Sun L, Song C, Moreno BH, Hu-Lieskovan S, Berent-Maoz B, Pang J, Chmielowski B, Cherry G, Seja E, Lomeli S, Kong X, Kelley MC, Sosman JA, Johnson DB, Ribas A, Lo RS. Genomic and Transcriptomic Features of Response to Anti-PD-1 Therapy in Metastatic Melanoma. Cell. 2016 Mar 24;165(1):35-44. doi: 10.1016/j.cell.2016.02.065. Epub 2016 Mar 17. PMID 26997480
- [Background] Hugo W, Zaretsky JM, Sun L, Song C, Moreno BH, Hu-Lieskovan S, Berent-Maoz B, Pang J, Chmielowski B, Cherry G, Seja E, Lomeli S, Kong X, Kelley MC, Sosman JA, Johnson DB, Ribas A, Lo RS. Genomic and Transcriptomic Features of Response to Anti-PD-1 Therapy in Metastatic Melanoma. Cell. 2017 Jan 26;168(3):542. doi: 10.1016/j.cell.2017.01.010. No abstract available. PMID 28129544
- [Background] Jones SJ, Laskin J, Li YY, Griffith OL, An J, Bilenky M, Butterfield YS, Cezard T, Chuah E, Corbett R, Fejes AP, Griffith M, Yee J, Martin M, Mayo M, Melnyk N, Morin RD, Pugh TJ, Severson T, Shah SP, Sutcliffe M, Tam A, Terry J, Thiessen N, Thomson T, Varhol R, Zeng T, Zhao Y, Moore RA, Huntsman DG, Birol I, Hirst M, Holt RA, Marra MA. Evolution of an adenocarcinoma in response to selection by targeted kinase inhibitors. Genome Biol. 2010;11(8):R82. doi: 10.1186/gb-2010-11-8-r82. Epub 2010 Aug 9. PMID 20696054
- [Background] Laskin J, Jones S, Aparicio S, Chia S, Ch'ng C, Deyell R, Eirew P, Fok A, Gelmon K, Ho C, Huntsman D, Jones M, Kasaian K, Karsan A, Leelakumari S, Li Y, Lim H, Ma Y, Mar C, Martin M, Moore R, Mungall A, Mungall K, Pleasance E, Rassekh SR, Renouf D, Shen Y, Schein J, Schrader K, Sun S, Tinker A, Zhao E, Yip S, Marra MA. Lessons learned from the application of whole-genome analysis to the treatment of patients with advanced cancers. Cold Spring Harb Mol Case Stud. 2015 Oct;1(1):a000570. doi: 10.1101/mcs.a000570. PMID 27148575
- [Background] Le DT, Uram JN, Wang H, Bartlett BR, Kemberling H, Eyring AD, Skora AD, Luber BS, Azad NS, Laheru D, Biedrzycki B, Donehower RC, Zaheer A, Fisher GA, Crocenzi TS, Lee JJ, Duffy SM, Goldberg RM, de la Chapelle A, Koshiji M, Bhaijee F, Huebner T, Hruban RH, Wood LD, Cuka N, Pardoll DM, Papadopoulos N, Kinzler KW, Zhou S, Cornish TC, Taube JM, Anders RA, Eshleman JR, Vogelstein B, Diaz LA Jr. PD-1 Blockade in Tumors with Mismatch-Repair Deficiency. N Engl J Med. 2015 Jun 25;372(26):2509-20. doi: 10.1056/NEJMoa1500596. Epub 2015 May 30. PMID 26028255
- [Background] Miao D, Margolis CA, Gao W, Voss MH, Li W, Martini DJ, Norton C, Bosse D, Wankowicz SM, Cullen D, Horak C, Wind-Rotolo M, Tracy A, Giannakis M, Hodi FS, Drake CG, Ball MW, Allaf ME, Snyder A, Hellmann MD, Ho T, Motzer RJ, Signoretti S, Kaelin WG Jr, Choueiri TK, Van Allen EM. Genomic correlates of response to immune checkpoint therapies in clear cell renal cell carcinoma. Science. 2018 Feb 16;359(6377):801-806. doi: 10.1126/science.aan5951. Epub 2018 Jan 4. PMID 29301960
- [Background] Newman AM, Liu CL, Green MR, Gentles AJ, Feng W, Xu Y, Hoang CD, Diehn M, Alizadeh AA. Robust enumeration of cell subsets from tissue expression profiles. Nat Methods. 2015 May;12(5):453-7. doi: 10.1038/nmeth.3337. Epub 2015 Mar 30. PMID 25822800
- [Background] Nielsen M, Andreatta M. NetMHCpan-3.0; improved prediction of binding to MHC class I molecules integrating information from multiple receptor and peptide length datasets. Genome Med. 2016 Mar 30;8(1):33. doi: 10.1186/s13073-016-0288-x. PMID 27029192
- [Background] Ock CY, Hwang JE, Keam B, Kim SB, Shim JJ, Jang HJ, Park S, Sohn BH, Cha M, Ajani JA, Kopetz S, Lee KW, Kim TM, Heo DS, Lee JS. Genomic landscape associated with potential response to anti-CTLA-4 treatment in cancers. Nat Commun. 2017 Oct 19;8(1):1050. doi: 10.1038/s41467-017-01018-0. PMID 29051489
- [Background] Palena C, Polev DE, Tsang KY, Fernando RI, Litzinger M, Krukovskaya LL, Baranova AV, Kozlov AP, Schlom J. The human T-box mesodermal transcription factor Brachyury is a candidate target for T-cell-mediated cancer immunotherapy. Clin Cancer Res. 2007 Apr 15;13(8):2471-8. doi: 10.1158/1078-0432.CCR-06-2353. PMID 17438107
- [Background] Panda A, Betigeri A, Subramanian K, Ross JS, Pavlick DC, Ali S, Markowski P, Silk A, Kaufman HL, Lattime E, Mehnert JM, Sullivan R, Lovly CM, Sosman J, Johnson DB, Bhanot G, Ganesan S. Identifying a Clinically Applicable Mutational Burden Threshold as a Potential Biomarker of Response to Immune Checkpoint Therapy in Solid Tumors. JCO Precis Oncol. 2017;2017:PO.17.00146. doi: 10.1200/PO.17.00146. Epub 2017 Dec 7. PMID 29951597
- [Background] Panda A, de Cubas AA, Stein M, Riedlinger G, Kra J, Mayer T, Smith CC, Vincent BG, Serody JS, Beckermann KE, Ganesan S, Bhanot G, Rathmell WK. Endogenous retrovirus expression is associated with response to immune checkpoint blockade in clear cell renal cell carcinoma. JCI Insight. 2018 Aug 23;3(16):e121522. doi: 10.1172/jci.insight.121522. eCollection 2018 Aug 23. PMID 30135306
- [Background] Peng W, Chen JQ, Liu C, Malu S, Creasy C, Tetzlaff MT, Xu C, McKenzie JA, Zhang C, Liang X, Williams LJ, Deng W, Chen G, Mbofung R, Lazar AJ, Torres-Cabala CA, Cooper ZA, Chen PL, Tieu TN, Spranger S, Yu X, Bernatchez C, Forget MA, Haymaker C, Amaria R, McQuade JL, Glitza IC, Cascone T, Li HS, Kwong LN, Heffernan TP, Hu J, Bassett RL Jr, Bosenberg MW, Woodman SE, Overwijk WW, Lizee G, Roszik J, Gajewski TF, Wargo JA, Gershenwald JE, Radvanyi L, Davies MA, Hwu P. Loss of PTEN Promotes Resistance to T Cell-Mediated Immunotherapy. Cancer Discov. 2016 Feb;6(2):202-16. doi: 10.1158/2159-8290.CD-15-0283. Epub 2015 Dec 8. PMID 26645196
- [Background] Pereira C, Gimenez-Xavier P, Pros E, Pajares MJ, Moro M, Gomez A, Navarro A, Condom E, Moran S, Gomez-Lopez G, Grana O, Rubio-Camarillo M, Martinez-Marti A, Yokota J, Carretero J, Galbis JM, Nadal E, Pisano D, Sozzi G, Felip E, Montuenga LM, Roz L, Villanueva A, Sanchez-Cespedes M. Genomic Profiling of Patient-Derived Xenografts for Lung Cancer Identifies B2M Inactivation Impairing Immunorecognition. Clin Cancer Res. 2017 Jun 15;23(12):3203-3213. doi: 10.1158/1078-0432.CCR-16-1946. Epub 2017 Mar 16. PMID 28302866
- [Background] Reisle C, Mungall KL, Choo C, Paulino D, Bleile DW, Muhammadzadeh A, Mungall AJ, Moore RA, Shlafman I, Coope R, Pleasance S, Ma Y, Jones SJM. MAVIS: merging, annotation, validation, and illustration of structural variants. Bioinformatics. 2019 Feb 1;35(3):515-517. doi: 10.1093/bioinformatics/bty621. PMID 30016509
- [Background] Roberts CW, Orkin SH. The SWI/SNF complex--chromatin and cancer. Nat Rev Cancer. 2004 Feb;4(2):133-42. doi: 10.1038/nrc1273. No abstract available. PMID 14964309
- [Background] Rowe HM, Trono D. Dynamic control of endogenous retroviruses during development. Virology. 2011 Mar 15;411(2):273-87. doi: 10.1016/j.virol.2010.12.007. Epub 2011 Jan 20. PMID 21251689
- [Background] Saunders CT, Wong WS, Swamy S, Becq J, Murray LJ, Cheetham RK. Strelka: accurate somatic small-variant calling from sequenced tumor-normal sample pairs. Bioinformatics. 2012 Jul 15;28(14):1811-7. doi: 10.1093/bioinformatics/bts271. Epub 2012 May 10. PMID 22581179
- [Background] Seymour L, Bogaerts J, Perrone A, Ford R, Schwartz LH, Mandrekar S, Lin NU, Litiere S, Dancey J, Chen A, Hodi FS, Therasse P, Hoekstra OS, Shankar LK, Wolchok JD, Ballinger M, Caramella C, de Vries EGE; RECIST working group. iRECIST: guidelines for response criteria for use in trials testing immunotherapeutics. Lancet Oncol. 2017 Mar;18(3):e143-e152. doi: 10.1016/S1470-2045(17)30074-8. Epub 2017 Mar 2. PMID 28271869
- [Background] Shen J, Ju Z, Zhao W, Wang L, Peng Y, Ge Z, Nagel ZD, Zou J, Wang C, Kapoor P, Ma X, Ma D, Liang J, Song S, Liu J, Samson LD, Ajani JA, Li GM, Liang H, Shen X, Mills GB, Peng G. ARID1A deficiency promotes mutability and potentiates therapeutic antitumor immunity unleashed by immune checkpoint blockade. Nat Med. 2018 May;24(5):556-562. doi: 10.1038/s41591-018-0012-z. Epub 2018 May 7. PMID 29736026
- [Background] Smart AC, Margolis CA, Pimentel H, He MX, Miao D, Adeegbe D, Fugmann T, Wong KK, Van Allen EM. Intron retention is a source of neoepitopes in cancer. Nat Biotechnol. 2018 Dec;36(11):1056-1058. doi: 10.1038/nbt.4239. Epub 2018 Aug 16. PMID 30114007
- [Background] Solovyov A, Vabret N, Arora KS, Snyder A, Funt SA, Bajorin DF, Rosenberg JE, Bhardwaj N, Ting DT, Greenbaum BD. Global Cancer Transcriptome Quantifies Repeat Element Polarization between Immunotherapy Responsive and T Cell Suppressive Classes. Cell Rep. 2018 Apr 10;23(2):512-521. doi: 10.1016/j.celrep.2018.03.042. PMID 29642008
- [Background] Strick R, Strissel PL, Baylin SB, Chiappinelli KB. Unraveling the molecular pathways of DNA-methylation inhibitors: human endogenous retroviruses induce the innate immune response in tumors. Oncoimmunology. 2015 Dec 29;5(5):e1122160. doi: 10.1080/2162402X.2015.1122160. eCollection 2016 May. PMID 27467919
- [Background] Szolek A, Schubert B, Mohr C, Sturm M, Feldhahn M, Kohlbacher O. OptiType: precision HLA typing from next-generation sequencing data. Bioinformatics. 2014 Dec 1;30(23):3310-6. doi: 10.1093/bioinformatics/btu548. Epub 2014 Aug 20. PMID 25143287
- [Background] Tumeh PC, Harview CL, Yearley JH, Shintaku IP, Taylor EJ, Robert L, Chmielowski B, Spasic M, Henry G, Ciobanu V, West AN, Carmona M, Kivork C, Seja E, Cherry G, Gutierrez AJ, Grogan TR, Mateus C, Tomasic G, Glaspy JA, Emerson RO, Robins H, Pierce RH, Elashoff DA, Robert C, Ribas A. PD-1 blockade induces responses by inhibiting adaptive immune resistance. Nature. 2014 Nov 27;515(7528):568-71. doi: 10.1038/nature13954. PMID 25428505
- [Background] Van Allen EM, Miao D, Schilling B, Shukla SA, Blank C, Zimmer L, Sucker A, Hillen U, Foppen MHG, Goldinger SM, Utikal J, Hassel JC, Weide B, Kaehler KC, Loquai C, Mohr P, Gutzmer R, Dummer R, Gabriel S, Wu CJ, Schadendorf D, Garraway LA. Genomic correlates of response to CTLA-4 blockade in metastatic melanoma. Science. 2015 Oct 9;350(6257):207-211. doi: 10.1126/science.aad0095. Epub 2015 Sep 10. PMID 26359337
- [Background] Vigneron N. Human Tumor Antigens and Cancer Immunotherapy. Biomed Res Int. 2015;2015:948501. doi: 10.1155/2015/948501. Epub 2015 Jun 16. PMID 26161423
- [Background] Warren RL, Choe G, Freeman DJ, Castellarin M, Munro S, Moore R, Holt RA. Derivation of HLA types from shotgun sequence datasets. Genome Med. 2012 Dec 10;4(12):95. doi: 10.1186/gm396. eCollection 2012. PMID 23228053
- [Background] Yang W, Lee KW, Srivastava RM, Kuo F, Krishna C, Chowell D, Makarov V, Hoen D, Dalin MG, Wexler L, Ghossein R, Katabi N, Nadeem Z, Cohen MA, Tian SK, Robine N, Arora K, Geiger H, Agius P, Bouvier N, Huberman K, Vanness K, Havel JJ, Sims JS, Samstein RM, Mandal R, Tepe J, Ganly I, Ho AL, Riaz N, Wong RJ, Shukla N, Chan TA, Morris LGT. Immunogenic neoantigens derived from gene fusions stimulate T cell responses. Nat Med. 2019 May;25(5):767-775. doi: 10.1038/s41591-019-0434-2. Epub 2019 Apr 22. PMID 31011208